CLINICAL TRIAL: NCT06271720
Title: Impact of Visceral Manipulation Versus Integrated Neuromuscular Inhibition Technique in Shoulder Impingement Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noha Elserty (Other)
Responsible Party: Sponsor-Investigator, Noha Elserty, Assistant professor, Egyptian Chinese University
Organization: Egyptian Chinese University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: faculty of physical therapy
Record Dates: First submitted 2024-01-19; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visceral manipulation (Active Comparator): Palpation will be applied and the pressure will directly to the skin, into the direction of restriction just until resistance (tissue barrier) is felt. Once found, the collagenous barrier will be engaged for 90 to 120 seconds for each technique without sliding over the skin or forcing the tissue until the fascia complex starts to yield and a sensation of softening is achieved.
  Interventions: Other: visceral manipulation
- integrated neuromuscular inhibition (Active Comparator): The practitioner first identifies TrPs to be treated within the upper trapezius muscle. The subjects will be placed in a supine position. Their arm will be positioned in slight shoulder abduction with the elbow bent and their hand resting on their stomach. Using a pincer grasp, the practitioner will move throughout the fibers of the upper trapezius and make note of any active TrPs. Once the TrPs were identified, treatment began. The first technique applied will be ischemic compression. The therapist again utilized a pincer grasp, placing the thumb and index finger over the active TrP. Slow, increasing levels of pressure will be applied until the tissue resistance barrier is identified. The pressure will be maintained until a release of the tissue barrier is felt. At that time, pressure will again be applied until a new barrier is felt. This process will be repeated until tension or tenderness is unable to be identified or 90 seconds have elapsed.
  Interventions: Other: integrated neuromuscular inhibition

INTERVENTIONS:
Other: visceral manipulation — visceral manipulation: A palpation technique will be applied till the barrier is felt and it will be applied until release is felt.
  integrated neuromuscular inhibition: ischemic compression will be applied to trigger point of upper trapezius
  Arms: visceral manipulation
Other: integrated neuromuscular inhibition — It involves applying direct sustained digital pressure to the TrP with sufficient force over dedicated time duration, to slow down the blood supply and relieve the tension within the involved muscle. The pressure is gradually applied, maintained and the gradually released
  Arms: integrated neuromuscular inhibition

SUMMARY:
This study will be conducted To evaluate the effect of Visceral Manipulation versus Integrated Neuromuscular Inhibition Technique on the upper fiber of trapezius on pain intensity, pain threshold, shoulder range of motion, and function in shoulder impingement syndrome

DETAILED DESCRIPTION:
HYPOTHESES

It will be hypothesized that:

1. There will be no statistically significant effect of Visceral Manipulation on the upper fiber of the trapezius on pain intensity, pain threshold, shoulder range of motion, or function in shoulder impingement syndrome
2. There will be no statistically significant effect of the Integrated Neuromuscular Inhibition Technique on the upper fiber of the trapezius on pain intensity, pain threshold, shoulder range of motion, or function in shoulder impingement syndrome.
3. There will be no statistically significant difference in the effect of visceral manipulation versus the integrated neuromuscular inhibition technique on the upper fiber of the trapezius on pain intensity, pain threshold, shoulder range of motion, and function in shoulder impingement syndrome.

This study will be conducted to answer the following questions:

Is there an effect of Visceral Manipulation versus Integrated Neuromuscular Inhibition Technique on the upper fiber of the trapezius on pain intensity, pain threshold, shoulder range of motion, and function in shoulder impingement syndrome?

ELIGIBILITY:
Inclusion Criteria:

* -active myofascial trigger points in the upper trapezius muscle, and chronic Pain lasting more than 12 weeks
* BMI between 25 and 30 Kg/m².

Exclusion Criteria:

* a previous fracture in the cervical spine or shoulder surgery
* acute inflammatory condition.
* Malignant tumor.
* Multiple osteophytes.
* Cervical posture abnormalities.
* Osteoporosis.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
pain intensity | pre treatment and after 4 weeks
  pain intensity will be measured by a visual analog scale, the scale is marked from 0 to 10 while 0 represents no pain and 10 represents intolerable pain
pain pressure threshold | pre treatment and after 4 weeks
  pressure threshold measured by pressure algometer
shoulder range of motion | pre treatment and after 4 weeks
  shoulder flexion and abduction range of motion will be measured by inclinometer
shoulder functional level | pre treatment and after 4 weeks
  The functional level of the shoulder will be measured by shoulder pain and disability index. the index consists of subscales that measure how much shoulder pain interferes with the functional activity of daily living